CLINICAL TRIAL: NCT06113848
Title: Feasibility and Efficacy of Intra- Arterial TNK and Albumin as an Adjunct to Thrombectomy for Acute Stroke
Brief Title: Adjunctive Use of Intra-Arterial TNK and Albumin Following Thrombectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJHH-2023-wm16
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Albumin; TNK; No-reflow; Endovascular Therapy; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Albumins; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intra-Arterial TNK and Albumin (Active Comparator)
  Interventions: Drug: Intra-Arterial TNK and Albumin
- Intra-Arterial TNK (Active Comparator)
  Interventions: Drug: Intra-Arterial TNK
- Intra-Arterial Albumin (Active Comparator)
  Interventions: Drug: Intra-Arterial Albumin
- sham (Sham Comparator)
  Interventions: Other: sham

INTERVENTIONS:
Drug: Intra-Arterial TNK and Albumin — The study population was divided into four groups, one of which had intra-arterial TNK and albumin.
  Arms: Intra-Arterial TNK and Albumin
Drug: Intra-Arterial TNK — The study population was divided into four groups, one of which had intra-arterial TNK .
  Arms: Intra-Arterial TNK
Drug: Intra-Arterial Albumin — The study population was divided into four groups, one of which had intra-arterial albumin.
  Arms: Intra-Arterial Albumin
Other: sham — The study population was divided into four groups, one of which had no intra-arterial TNK and albumin.
  Arms: sham

SUMMARY:
The purpose of this study is to investigate the feasibility and efficacy of intra-arterial TNK and albumin for patients with acute ischemic stroke after successful thrombectomy and whether there is a synergistic effect between TNK and albumin.

DETAILED DESCRIPTION:
Endovascular therapy is the first-line treatment for acute ischemic stroke with large vessel occlusion. However, many studies have shown that, even with successful recanalization, about half of patients do not achieve functional independence. This phenomenon is called futile recanalization, which is partly attributed to brain no-reflow (microcirculation reperfusion failure despite recanalization of the occluded large artery). The mechanisms of brain no-reflow phenomenon include inflammation, micro thrombosis, aggregation platelets and red blood cells, and pericyte contraction.

Albumin, the most copious plasma protein synthesized primarily in the liver, possesses various biochemical properties, including anti-inflammatory, inhibiting platelet aggregation and micro thrombosis formation, and increasing microvascular perfusion. All of these properties are directed toward the mechanisms of no-reflow production, so albumin may inhibit no-reflow to improve the prognosis of stroke patients. TNK is a new generation thrombolytic agent that inhibits thrombosis, improves microcirculatory perfusion, and may inhibit no-reflow. These functions of TNK are similar to those of albumin, and the two also can reduce infraction volume and cerebral edema, and improve of behavioral function. In this study, we plan to determine the feasibility and efficacy of intra-arterial TNK and albumin for stroke patients undergoing successful mechanical thrombectomy and whether there is a synergistic effect between TNK and albumin.

ELIGIBILITY:
Inclusion criteria:

1. AIS patients with large vessel occlusion;
2. Age between 18 and 80 years;
3. Baseline NIHSS score ≥ 6; 4 .Successful recanalization after thrombectomy (mTICI grades ≥ 2b);

5. ASPECTS score ≥ 6 on CT; 6. First episode or previous episode without significant sequelae (mRS ≤ 2); 7. Time from onset to femoral artery puncture ≤ 24 hours; 8. Written informed consent provided by the patients or their legal relatives.

Exclusion criteria:

1. Upon admission, the patient's medical history and physical examination revealed manifestations indicative of congestive heart failure (CHF), such as jugular venous distention, the presence of a third heart sound, resting tachycardia at a rate of 100 beats per minute attributable to heart failure, hepatomegaly, and/or lower extremity edema attributable to heart failure or of unknown etiology;
2. History of acute myocardial infarction within the preceding 3 months;
3. The patient's medical history, electrocardiogram findings upon admission, or physical examination indicated the presence of second- or third-degree heart block or any arrhythmia associated with hemodynamic instability, as determined by the investigator's assessment;
4. Acute or chronic renal failure with serum creatinine levels exceeding 2.0 mg/dL;
5. Severe anemia characterized by a hematocrit below 32%;
6. Computed tomography findings upon admission indicating the presence of any form of hemorrhage;
7. Pregnancy status;
8. Previous history of allergic reactions to albumin administration or TNK administration;
9. Elevated blood pressure exceeding 185/110 mmHg when investigating the use of albumin administration or TNK administration;
10. Presence of other potentially life-threatening medical conditions;
11. Individuals with current chronic lung diseases, such as chronic obstructive pulmonary disease, bronchiectasis, or any other lung disorder that significantly impairs daily activities;
12. Individuals with known allergies to albumin or TNK;
13. Patients with reocclusion within 24 hours;
14. Clinical suspicion of aortic coarctation、 bacterial embolism and infective endocarditis;
15. Patients with a history of coagulation disorders and systemic bleeding tendencies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-09-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major response | 7 days after initiation of TNK or albumin intra-arterially
  Major response is any of the following:
  1. Any forms of intracranial hemorrhage;
  2. Pulmonary edema;
  3. Heart failure;
  4. Skin itching, dyspnea and other allergic reactions;
  5. Death of any causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No